CLINICAL TRIAL: NCT02577666
Title: Evaluation of EBT With Young, Substance Abusing Homeless Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Natasha Slesnick, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014B0348; R01DA023062 (NIH)
Record Dates: First submitted 2015-10-10; First posted 2015-10-16 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ecologically-Based Therapy + TAU (Experimental): receives Ecologically-Based Therapy which includes the Community Reinforcement Approach, Strengths-Based Case Management (6 months) and rental assistance for housing (3 months) + TAU
  Interventions: Behavioral: Ecologically Based Therapy; Behavioral: Treatment as Usual
- Housing Only + TAU (Experimental): receives 3 months of rental assistance for housing only + TAU
  Interventions: Behavioral: Housing Only; Behavioral: Treatment as Usual
- treatment as usual (TAU) (Other): receives usual treatments/interventions (TAU) within in the community
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Ecologically Based Therapy — 6 months of community reinforcement approach and case management, 3 months of rental assistance for housing
  Arms: Ecologically-Based Therapy + TAU
Behavioral: Housing Only — receives 3 months of project supported rental assistance
  Arms: Housing Only + TAU
Behavioral: Treatment as Usual — receives services as normally offered within the community

SUMMARY:
A dearth of information is available regarding how best to intervene with substance use disordered homeless mothers and their young children. This proposal follows from the promising findings of a rigorously developed ecologically based treatment that offers a comprehensive intervention for the multiple needs of this vulnerable population. Such research attention is needed in order to effectively intervene in the substance use, HIV risk, mental/physical health and homeless trajectory of these women and their young children. Further, if successful, this intervention may be transportable to communities without crisis shelters and to homeless mothers who do not access shelter or residential treatment services.

DETAILED DESCRIPTION:
Homeless mothers with young children in their care contend with high rates of substance use, HIV risk, physical and mental health problems and parenting stress. These struggles are in addition to homelessness and meeting the basic needs of themselves and their children. However, a very limited number of studies have examined mother and child outcomes associated with housing and supportive services. Even with increased focus on those experiencing homelessness, the number of homeless families continues to rise, with the demand for temporary shelter so high that many cities are unable to meet the needs of these families. A comprehensive intervention that can be offered outside the shelter setting may offer greater reach to those experiencing homelessness who do not make it in to the shelter system, and for those communities that do not have shelters available. Among the young homeless, those under age 25, research documents that the majority (70%) have never used shelter services. Research attention towards identifying efficacious interventions for this population which address the multiple needs of these families is thus considered an important focus. The proposed intervention (Ecologically-Based Treatment, EBT) includes housing and supportive services and utilizes an ecological systems approach as the theoretical base. It was rigorously developed in a Stage 1 treatment development study with substance use disordered homeless mothers who were engaged through a crisis shelter. EBT showed several outcomes superior to shelter services and is therefore considered a good fit for a population who avoids the shelter but is in great need of housing and support services. Two hundred forty (N = 240) substance use disordered homeless young women between the ages of 18 to 24 years with a biological child under the age of 6 years in their care will be randomly assigned to one of three conditions:

1. housing and support services (EBT) + Treatment as Usual (TAU) (N = 80),
2. housing only (HO) + TAU (N = 80), or
3. TAU only (N=80).

EBT includes 6 months of supportive services (case management, HIV prevention and the Community Reinforcement Approach) in addition to 3 months of rental assistance. HO includes 3 months of rental assistance, but without supportive services. TAU is usual services offered by a homeless youth drop-in center. Participants will be re-assessed at 3, 6, 9 and 12 months post-baseline. Theoretically derived mediators of change as well as a formal economic evaluation will offer important policy implications. Since homeless substance use disordered mothers and their children are at increased risk for a variety of adverse outcomes, the intervention may produce substantial health-care benefits to their families and society at large.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-24 years
* meets McKinney-Vento definition of homeless
* has physical custody of child under the age of 7
* meets DSM5 criteria for alcohol/drug use disorder

Exclusion Criteria:

* Evidence of unremitted psychosis or other condition which would impair mother's ability to understand or participate in the intervention or consent to the research

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-02; Primary Completion 2018-10 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in substance use frequency | 12 months
  frequency of substance use is measured at baseline, 3, 6, 9 and 12-months post-baseline

SECONDARY OUTCOMES:
change in stable housing | 12 months
  number of days in own apartment paying rent is measured at baseline, 3, 6, 9 and 12 months post-baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Department of Human Development and Family Science, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT02577666/ICF_000.pdf